CLINICAL TRIAL: NCT04881461
Title: A Randomised, Parallel-group, Double-blind, Placebo-controlled Phase III Trial Assessing the Efficacy and Safety of 5-grass Mix SLIT-drops in Adults With Grass Pollen-induced Rhinoconjunctivitis
Brief Title: A Study in Adults With Grass Pollen-induced Rhinoconjunctivitis
Acronym: Rhapsody
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ALK-Abelló A/S (Industry)
Collaborators: Syneos Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SU-G-01; 2020-000455-12 (EudraCT Number)
Record Dates: First submitted 2021-03-18; First posted 2021-05-11 (Actual); Results first posted 2024-12-16 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Allergy
Keywords: Allergic rhinoconjunctivitis; Adults; Grass
MeSH Terms: conditions — Hypersensitivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Glycerol, carbonate, sodium chloride One single-dose container (0.5 ml) once daily
  Interventions: Drug: Placebo
- 5-grass mix SLIT-drops (Experimental): Grass mix sublingual allergy immunotherapy drops One single-dose container (0.5 ml) once daily. 50 SRU/day for five consecutive days followed by 150 SRU/day for five additional consecutive days. Maintenance: 300 SRU/day from day 11.
  Interventions: Drug: 5-grass mix SLIT-drops

INTERVENTIONS:
Drug: 5-grass mix SLIT-drops — Sublingual allergy immunotherapy drops, for daily administration
  Other Names: SLIToneULTRA
  Arms: 5-grass mix SLIT-drops
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a 2 year clinical study to compare 5-grass mix SLIT-drops with placebo in relieving grass pollen-induced rhinoconjunctivitis symptoms and in use of symptom-relieving medication during the second grass pollen season (peak grass pollen season, PGPS)

The study will collect health-related quality of life data in the groups treated with 5-grass mix SLIT-drops or with placebo during the first and second PGPS.

The trial medication used is already approved to treat allergic rhinitis caused by grass pollen in adults in several countries.

DETAILED DESCRIPTION:
This trial is a 2 year, parallel-group, double-blind, placebo-controlled phase III trial to evaluate efficacy and safety of the 5-grass mix SLIT-drops in adults with grass pollen-induced rhinoconjunctivitis with or without asthma. Approximately 440 adults will be enrolled in the trial and will receive the 5-grass mix SLIT-drops or placebo. The trial is conducted in several European countries.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged ≥18 years on the day informed consent is obtained
2. A clinical history of grass pollen-induced allergic rhinoconjunctivitis for two years or more with or without asthma
3. A clinical history of severe allergic rhinoconjunctivitis symptoms (interfering with usual daily activities or sleep) induced by grass pollen, which remain troublesome despite symptomatic treatment with antihistamines, nasal steroids or eye drops during the previous grass pollen season
4. Positive specific immunoglobulin E (IgE) (defined as ≥class 2, ≥0.70 kU/l) against grass: Phleum pratense
5. Positive skin prick test to Phleum pratense at screening

Exclusion Criteria:

1. Has a clinically relevant history of symptomatic seasonal and/or perennial allergic rhinoconjunctivitis and/or asthma caused by an allergen other than grass pollen, to which the subject is exposed, which could potentially overlap with the efficacy assessment periods
2. Within the last 3 months before the randomisation visit, has had an occurrence of any clinical deterioration of asthma that resulted in emergency treatment, hospitalisation, or treatment with systemic corticosteroids
3. SLIT treatment with any grass pollen AIT for more than 1 month within the last 5 years. In addition, any SLIT treatment with grass pollen AIT within the previous 12 months
4. SCIT treatment with any grass AIT reaching the maintenance dose within the last 5 years. In addition, any SCIT treatment with grass AIT within the previous 12 months
5. Ongoing treatment with any allergy immunotherapy product
6. Uncontrolled or severe asthma requiring daily use of more than 800 mcg budesonide or equivalent at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 445 (Actual)
Dates: Start 2021-05-10 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-09-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laurent Guilleminault, MD, Principal Investigator — CHU Hôpital Larrey
Locations (48):
- Czechia (9):
  - Fakultni Nemocnice u Sv. Anny - FNUSA, Brno
  - Ambulance alergologie a klinicke imunologie - Ceske Budejovice, České Budějovice
  - Alergopraktik s.r.o., Jablonec nad Nisou
  - Allergology Jihlava, Jihlava
  - Alergologicka Ambulance - Liberec, Liberec
  - Alergomyšl s.r.o, Litomyšl
  - Acredula Benedicta s.r.o., Pardubice
  - KASMED s.r.o., Tábor
  - MUJ ALERGOLOG s.r.o., Trutnov
- North Estonia Medical Centre Foundation, Tallinn, Estonia
- France (9):
  - Hopital Privé de la Loire, Loiré, Saint-Étienne
  - Cabinet medical, Fenouillet
  - Cabinet medical, Hyères
  - Cabinet medical, Joué-lès-Tours
  - Cabinet medical, Paris
  - Cabinet médical, Rezé
  - Cabinet medical, Saint-Quentin
  - Nouvel Hopital Civil, Strasbourg
  - CHU Hôpital Larrey, Toulouse
- Latvia (6):
  - M & M Centrs LTD, Ādaži
  - Balvu and Gulbenes hospital union, Balvi
  - Daugavpils Regional hospital, Outpatient clinic, Daugavpils
  - Vevere Viktorija - Doctor's Practice in Pneumology and Allergology, Rēzekne
  - Ozola Inese - Family doctor's practice, Riga
  - The Centre of Investigation and Treatment of Allergic Diseases, Riga
- Lithuania (8):
  - JSC Ausros Medicinos Centras, Kaunas
  - Hospital of Lithuanian University of Health Sciences Kauno klinikos, Kaunas
  - JSC Inlita, Klaipedos CTC, Klaipėda
  - JSC Seimos gydytojas, Vilnius
  - JSC Center of Innovative Allergology, Vilnius
  - JSC INLITA, Santaros CTC, Vilnius
  - Allergy Clinic JSC Perspektyvos, Vilnius
  - JSC Center for Diagnosis and Treatment of Allergic Diseases, Vilnius
- Poland (15):
  - Snzoz Alergologia Plus Ośrodek Diagnostyki i Terapii Uczuleń, Poznan, Greater Poland Voivodeship
  - Grażyna Pulka Centrum Medyczne ALL-MED, Krakow, Lesser Poland Voivodeship
  - Alergo-Med Specjalistycza Przychodnia Lekarska Sp. zo.o., Tarnów, Maopolskie
  - Indywidualna Specjalistyczna Praktyka Lekarska Anna Latos, Kielce
  - Centrum Usług Medycznych Dyga-Med, Krakow
  - Grażyna Jasieniak-Pinis ATOPIA NZOZ Poradnie Specjalistyczne, Krakow
  - Barbara Rewerska Diamond Clinic, Krakow
  - Specjalistyczna Przychodnia Alergologiczna Centrum Alergologii, Lublin
  - Centrum Alergologii T.Hofman Sp. Z o.o., Poznan
  - Snzoz Imedica, Poznan
  - Prywatny Gabinet Lekarski Małgorzata Pawlukiewicz, Rzeszów
  - Gabinet Lekarski Bozena Kubicka-Kozik, Tomaszów Mazowiecki
  - ALL-MED. Specjalistyczna Opieka Medyczna. Medyczny Instytut Badawczy. Marek Jutel., Wroclaw
  - NZOZ Centrum Usług Medycznych Proximum Sp. z o.o., Wroclaw
  - Lekarze Specjaliści Malolepszy i Partnerzy, Wroclaw

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 445 participants were randomized and treated. Participants were recruited from 45 sites in 6 countries (Czechia, Estonia, France, Latvia, Lithuania, and Poland).
Groups:
- Placebo: Daily placebo sublingual immunotherapy drops (Placebo SLIT-drops) plus rhinoconjunctivitis rescue medication as needed.
- 5-grass Mix SLIT-drops: Daily grass sublingual immunotherapy drops (5-grass mix SLIT-drops) plus rhinoconjunctivitis rescue medication as needed.
Period: Overall Study
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Started (Randomized and treated) | 223 | 222
Completed (Completed trial) | 196 | 193
Not Completed | 27 | 29
Not completed — Adverse Event | 2 | 4
Not completed — Withdrawal by Subject | 19 | 19
Not completed — Lost to Follow-up | 4 | 4
Not completed — Lack of Efficacy | 1 | 0
Not completed — Reason stated as "other" in CRF | 1 | 2

BASELINE CHARACTERISTICS:
Population: All randomized and treated participants
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 5-grass Mix SLIT-drops | Total
Number analyzed (Participants) | 223 | 222 | 445
Age, Continuous [Mean (Standard Deviation); unit: Years] | 33.0 (9.7) | 32.2 (10.1) | 32.6 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 105 | 95 | 200
  Male | 118 | 127 | 245
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 223 | 222 | 445
Region of Enrollment [Number; unit: participants]
  Czechia | 56 | 57 | 113
  Estonia | 2 | 0 | 2
  France | 6 | 7 | 13
  Latvia | 17 | 16 | 33
  Lithuania | 25 | 26 | 51
  Poland | 117 | 116 | 233
Ongoing asthma [Count of Participants; unit: Participants] | 63 | 59 | 122

OUTCOME MEASURES:

1. Primary Outcome: Average Daily Allergic Rhinoconjunctivitis Total Combined Score (TCS) During the 2nd Peak Grass Pollen Season (PGPS)
Description: The average daily TCS evaluates the treatment effect based on reduction in daily rhinoconjunctivitis symptoms and in use of symptom-relieving medication (on a scale from 0 to 38). Higher scores indicate more severe symptoms and/or more medication use. The endpoint is calculated as the average score of all reported daily values during the 2nd PGPS.
Time Frame: During the 2nd PGPS (14 days)
Population: Participants in the full analysis set.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Number analyzed (Participants) | 192 | 187
score on a scale | 7.10 (0.51) | 5.22 (0.42)
Statistical Analysis 1: Comparison: Placebo vs 5-grass Mix SLIT-drops; The null hypothesis was defined as "no difference in means between treatment arms". The endpoint analysis was based on a 5% significance level. The trial was designed to have 86% power for the primary endpoint using the primary (trial product) estimand; Test type: Superiority; p = 0.0036, Mixed Models Analysis — Adjusted P-value; Covariates in the model: treatment, season and their interaction, ongoing asthma status, and country and season interaction; Mean Difference (Final Values) = 1.88, 95% CI 2-sided [0.60 to 3.17] — Placebo vs 5-grass mix SLIT-drops

2. Secondary Outcome: Average Weekly Overall Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Score During the 2nd Peak Grass Pollen Season (PGPS)
Description: The RQLQ measures the rhinoconjunctivitis quality of life. The RQLQ contains 28 questions, each scored on a 7-point scale (0 = not impaired at all; 6 = severely impaired). The overall RQLQ score is a mean of the 28 questions. Higher scores indicate worse quality of life. The endpoint is calculated as the average score of all reported weekly values during the 2nd PGPS.
Time Frame: During the 2nd PGPS (14 days)
Population: Participants in the full analysis set.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Number analyzed (Participants) | 187 | 182
score on a scale | 1.04 (0.08) | 0.86 (0.08)
Statistical Analysis 1: Comparison: Placebo vs 5-grass Mix SLIT-drops; The null hypothesis was defined as "no difference in means between treatment arms". The endpoint analysis was based on a 5% significance level. The trial was designed to have 95% power for this key secondary endpoint using the primary (trial product) estimand; Test type: Superiority; p = 0.1111, Mixed Models Analysis — Adjusted P-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.17, 95% CI 2-sided [-0.04 to 0.39] — Placebo vs 5-grass mix SLIT-drops

3. Secondary Outcome: Average Daily Allergic Rhinoconjunctivitis Total Combined Score (TCS) During the 1st Peak Grass Pollen Season (PGPS)
Description: The average daily TCS evaluates the treatment effect based on reduction in daily rhinoconjunctivitis symptoms and in use of symptom-relieving medication (on a scale from 0 to 38). Higher scores indicate more severe symptoms and/or more medication use. The endpoint is calculated as the average score of all reported daily values during the 1st PGPS.
Time Frame: During the 1st PGPS (14 days)
Population: Participants in the full analysis set.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Number analyzed (Participants) | 207 | 203
score on a scale | 8.10 (0.54) | 6.76 (0.42)
Statistical Analysis 1: Comparison: Placebo vs 5-grass Mix SLIT-drops; The null hypothesis was defined as "no difference in means between treatment arms". The analysis was based on a 5% significance level. The endpoint was analysed using primary (trial product) estimand; Test type: Superiority; p = 0.0417, Mixed Models Analysis — Observed P-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.33, 95% CI 2-sided [-0.01 to 2.67] — Placebo vs 5-grass SLIT-drops

4. Secondary Outcome: Average Weekly Overall Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Score During the 1st Peak Grass Pollen Season (PGPS)
Description: The RQLQ measures the rhinoconjunctivitis quality of life. The RQLQ contains 28 questions, each scored on a 7-point scale (0 = not impaired at all; 6 = severely impaired). The overall RQLQ score is a mean of the 28 questions. Higher scores indicate worse quality of life. The endpoint is calculated as the average score of all reported weekly values during the 1st PGPS.
Time Frame: During the 1st PGPS (14 days)
Population: Participants in the full analysis set.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Number analyzed (Participants) | 205 | 197
score on a scale | 1.26 (0.09) | 1.19 (0.08)
Statistical Analysis 1: Comparison: Placebo vs 5-grass Mix SLIT-drops; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4984, Mixed Models Analysis — Observed P-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.08, 95% CI 2-sided [-0.15 to 0.30] — Placebo vs 5-grass SLIT drops

5. Secondary Outcome: Average Weekly Overall Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Score During the 1st Entire Grass Pollen Season (EGPS)
Description: The RQLQ measures the rhinoconjunctivitis quality of life. The RQLQ contains 28 questions, each scored on a 7-point scale (0 = not impaired at all; 6 = severely impaired). The overall RQLQ score is a mean of the 28 questions. Higher scores indicate worse quality of life. The endpoint is calculated as the average score of all reported weekly values during the 1st EGPS.
Time Frame: During the 1st EGPS (observed mean duration of approximately 8 weeks)
Population: Participants in the full analysis set.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Number analyzed (Participants) | 207 | 205
score on a scale | 1.16 (0.09) | 1.09 (0.08)
Statistical Analysis 1: Comparison: Placebo vs 5-grass Mix SLIT-drops; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4438, Mixed Models Analysis — Observed P-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.07, 95% CI 2-sided [-0.12 to 0.27] — Placebo vs 5-grass mix SLIT-drops

6. Secondary Outcome: Average Weekly Overall Rhinoconjunctivitis Quality of Life Questionnaire (RQLQ) Score During the 2nd Entire Grass Pollen Season (EGPS)
Description: The RQLQ measures the rhinoconjunctivitis quality of life. The RQLQ contains 28 questions, each scored on a 7-point scale (0 = not impaired at all; 6 = severely impaired). The overall RQLQ score is a mean of the 28 questions. Higher scores indicate worse quality of life. The endpoint is calculated as the average score of all reported weekly values during the 2nd EGPS.
Time Frame: During the 2nd EGPS (observed mean duration of approximately 9 weeks)
Population: Participants in the full analysis set.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Number analyzed (Participants) | 192 | 190
score on a scale | 1.03 (0.08) | 0.83 (0.07)
Statistical Analysis 1: Comparison: Placebo vs 5-grass Mix SLIT-drops; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0363, Mixed Models Analysis — Observed P-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.20, 95% CI 2-sided [0.01 to 0.38] — Placebo vs 5-grass mix SLIT-drops

7. Secondary Outcome: Average Daily Allergic Rhinoconjunctivitis Total Combined Score (TCS) During the 1st Entire Grass Pollen Season (EGPS)
Description: The average daily TCS evaluates the treatment effect based on reduction in daily rhinoconjunctivitis symptoms and in use of symptom-relieving medication (on a scale from 0 to 38). Higher scores indicate more severe symptoms and/or more medication use. The endpoint is calculated as the average score of all reported daily values during the 1st EGPS.
Time Frame: During the 1st EGPS (observed mean duration of approximately 8 weeks)
Population: Participants in the full analysis set.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Number analyzed (Participants) | 207 | 205
score on a scale | 7.42 (0.54) | 6.23 (0.45)
Statistical Analysis 1: Comparison: Placebo vs 5-grass Mix SLIT-drops; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0329, Mixed Models Analysis — Observed P-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.19, 95% CI 2-sided [0.06 to 2.31] — Placebo vs 5-grass mix SLIT drops

8. Secondary Outcome: Average Daily Allergic Rhinoconjunctivitis Total Combined Score (TCS) During the 2nd Entire Grass Pollen Season (EGPS)
Description: The average daily TCS evaluates the treatment effect based on reduction in daily rhinoconjunctivitis symptoms and in use of symptom-relieving medication (on a scale from 0 to 38). Higher scores indicate more severe symptoms and/or more medication use. The endpoint is calculated as the average score of all reported daily values during the 2nd EGPS.
Time Frame: During the 2nd EGPS (observed mean duration of approximately 9 weeks)
Population: Participants in the full analysis set.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Number analyzed (Participants) | 193 | 190
score on a scale | 6.58 (0.50) | 4.86 (0.43)
Statistical Analysis 1: Comparison: Placebo vs 5-grass Mix SLIT-drops; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0016, Mixed Models Analysis — Observed P-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.73, 95% CI 2-sided [0.66 to 2.79] — Placebo vs 5-grass mix SLIT-drops

9. Secondary Outcome: Average Allergic Rhinoconjunctivitis Daily Symptoms Score (DSS) During the 1st Peak Grass Pollen Season (PGPS)
Description: The average DSS evaluates the treatment effect based on reduction in daily rhinoconjunctivitis symptoms (on a scale from 0 to18). Higher scores indicate more severe symptoms. The endpoint is calculated as the average score of all reported daily values during the 1st PGPS.
Time Frame: During the 1st PGPS (14 days)
Population: Participants in the full analysis set.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Number analyzed (Participants) | 207 | 203
score on a scale | 4.08 (0.27) | 3.83 (0.23)
Statistical Analysis 1: Comparison: Placebo vs 5-grass Mix SLIT-drops; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4502, Mixed Models Analysis — Observed P-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.25, 95% CI 2-sided [-0.42 to 0.92] — Placebo vs 5-grass mix SLIT-drops

10. Secondary Outcome: Average Allergic Rhinoconjunctivitis Daily Symptoms Score (DSS) During the 2nd Peak Grass Pollen Season (PGPS)
Description: The average DSS evaluates the treatment effect based on reduction in daily rhinoconjunctivitis symptoms (on a scale from 0 to18). Higher scores indicate more severe symptoms. The endpoint is calculated as the average score of all reported daily values during the 2nd PGPS.
Time Frame: During the 2nd PGPS (14 days)
Population: Participants in the full analysis set.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Number analyzed (Participants) | 192 | 187
score on a scale | 3.64 (0.26) | 3.09 (0.25)
Statistical Analysis 1: Comparison: Placebo vs 5-grass Mix SLIT-drops; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.1177, Mixed Models Analysis — Observed P-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.55, 95% CI 2-sided [-0.14 to 1.23] — Placebo vs 5-grass mix SLIT-drops

11. Secondary Outcome: Average Allergic Rhinoconjunctivitis Daily Symptoms Score (DSS) During the 1st Entire Grass Pollen Season (EGPS)
Description: The average DSS evaluates the treatment effect based on reduction in daily rhinoconjunctivitis symptoms (on a scale from 0 to18). Higher scores indicate more severe symptoms. The endpoint is calculated as the average score of all reported daily values during the 1st EGPS.
Time Frame: During the 1st EGPS (observed mean duration of approximately 8 weeks)
Population: Participants in the full analysis set.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Number analyzed (Participants) | 207 | 205
score on a scale | 3.82 (0.24) | 3.61 (0.22)
Statistical Analysis 1: Comparison: Placebo vs 5-grass Mix SLIT-drops; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.4604, Mixed Models Analysis — Observed P-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.21, 95% CI 2-sided [-0.37 to 0.79] — Placebo vs 5-grass mix SLIT-drops

12. Secondary Outcome: Average Allergic Rhinoconjunctivitis Daily Symptoms Score (DSS) During the 2nd Entire Grass Pollen Season (EGPS)
Description: The average DSS evaluates the treatment effect based on reduction in daily rhinoconjunctivitis symptoms (on a scale from 0 to18). Higher scores indicate more severe symptoms. The endpoint is calculated as the average score of all reported daily values during the 2nd EGPS.
Time Frame: During the 2nd EGPS (observed mean duration of approximately 9 weeks)
Population: Participants in the full analysis set.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Number analyzed (Participants) | 193 | 190
score on a scale | 3.46 (0.23) | 2.89 (0.22)
Statistical Analysis 1: Comparison: Placebo vs 5-grass Mix SLIT-drops; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0549, Mixed Models Analysis — Observed P-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.57, 95% CI 2-sided [-0.01 to 1.15] — Placebo vs 5-grass mix SLIT-drops

13. Secondary Outcome: Average Allergic Rhinoconjunctivitis Daily Medication Score (DMS) During the 1st Peak Grass Pollen Season (PGPS)
Description: The average DMS evaluates the treatment effect based on reduction in daily use of rhinoconjunctivitis symptom-relieving medication (on a scale from 0 to 20). Higher scores indicate more medication use. The endpoint is calculated as the average score of all reported daily values during the 1st PGPS.
Time Frame: During the 1st PGPS (14 days)
Population: Participants in the full analysis set.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Number analyzed (Participants) | 207 | 203
units on a scale | 3.34 (0.34) | 2.23 (0.25)
Statistical Analysis 1: Comparison: Placebo vs 5-grass Mix SLIT-drops; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0049, Mixed Models Analysis — Observed P-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.12, 95% CI 2-sided [0.30 to 1.93] — Placebo vs 5-grass mix SLIT-drops

14. Secondary Outcome: Average Allergic Rhinoconjunctivitis Daily Medication Score (DMS) During the 2nd Peak Grass Pollen Season (PGPS)
Description: The average DMS evaluates the treatment effect based on reduction in daily use of rhinoconjunctivitis symptom-relieving medication (on a scale of 0 to 20). Higher scores indicate more medication use. The endpoint is calculated as the average score of all reported daily values during the 2nd PGPS.
Time Frame: During the 2nd PGPS (14 days)
Population: Participants in the full analysis set.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Number analyzed (Participants) | 192 | 187
score on a scale | 2.77 (0.30) | 1.52 (0.21)
Statistical Analysis 1: Comparison: Placebo vs 5-grass Mix SLIT-drops; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0004, Mixed Models Analysis — Observed P-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.24, 95% CI 2-sided [0.54 to 1.95] — Placebo vs 5-grass mix SLIT-drops

15. Secondary Outcome: Average Allergic Rhinoconjunctivitis Daily Medication Score (DMS) During the 1st Entire Grass Pollen Season (EGPS)
Description: The average DMS evaluates the treatment effect based on reduction in daily use of rhinoconjunctivitis symptom-relieving medication(on a scale from 0 to 20). Higher scores indicate more medication use. The endpoint is calculated as the average score of all reported daily values during the 1st EGPS.
Time Frame: During the 1st EGPS (observed mean duration of approximately 8 weeks)
Population: Participants in the full analysis set.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Number analyzed (Participants) | 207 | 205
score on a scale | 3.04 (0.35) | 2.10 (0.27)
Statistical Analysis 1: Comparison: Placebo vs 5-grass Mix SLIT-drops; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0054, Mixed Models Analysis — Observed P-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.94, 95% CI 2-sided [0.25 to 1.63] — Placebo vs 5-grass mix SLIT-drops

16. Secondary Outcome: Average Allergic Rhinoconjunctivitis Daily Medication Score (DMS) During the 2nd Entire Grass Pollen Season (EGPS)
Description: The average DMS evaluates the treatment effect based on reduction in daily use of rhinoconjunctivitis symptom-relieving medication (on a scale from 0 to 20). Higher scores indicate more medication use. The endpoint is calculated as the average score of all reported daily values during the 2nd EGPS.
Time Frame: During the 2nd EGPS (observed mean duration of approximately 9 weeks)
Population: Participants in the full analysis set.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 5-grass Mix SLIT-drops
Number analyzed (Participants) | 193 | 190
score on a scale | 2.62 (0.31) | 1.51 (0.23)
Statistical Analysis 1: Comparison: Placebo vs 5-grass Mix SLIT-drops; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.0002, Mixed Models Analysis — Observed P-value; [statistical method as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.11, 95% CI 2-sided [0.52 to 1.71] — Placebo vs 5-grass mix SLIT-drops

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) were collected from consent until the last follow-up phone contact with the participant (approximately 26 months of treatment). The displayed AEs were collected starting on/after time of first IMP administration and no later than 7 days after last IMP administration.
Description: All AEs starting on/after time of first IMP administration and no later than 7 days after last IMP administration are displayed. Both treatment-related and non-treatment-related AEs are displayed.
Arm/Group | Placebo | 5-grass Mix SLIT-drops
All-Cause Mortality (participants affected / at risk) | 0/223 | 0/222
Serious Adverse Events (participants affected / at risk) | 6/223 | 4/222
Other Adverse Events (participants affected / at risk) | 111/223 | 128/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=223) | 5-grass Mix SLIT-drops (N=222)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Gastrointestinal procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Choking (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Device breakage (Product Issues) | 1 (1) | 0 (0)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=223) | 5-grass Mix SLIT-drops (N=222)
COVID-19 (Infections and infestations) | 43 (50) | 41 (44)
Nasopharyngitis (Infections and infestations) | 43 (75) | 38 (67)
Viral infection (Infections and infestations) | 7 (8) | 14 (15)
Influenza (Infections and infestations) | 11 (13) | 12 (12)
Upper respiratory tract infection (Infections and infestations) | 15 (20) | 10 (19)
Bronchitis (Infections and infestations) | 14 (15) | 7 (9)
Pharyngitis (Infections and infestations) | 20 (25) | 4 (4)
Oral pruritus (Gastrointestinal disorders) | 11 (12) | 40 (49)
Oral discomfort (Gastrointestinal disorders) | 1 (1) | 15 (18)
Mouth swelling (Gastrointestinal disorders) | 0 (0) | 13 (15)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 16 (16)
Headache (Nervous system disorders) | 19 (30) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication can be made before the first multi-center publication. PI shall allow Sponsor (S) no less than 60 days to review publications and presentations. S can comment and require removal of confidential information. Upon S request, PI must delay the publication or presentation for 6 months to permit S to file a patent application or take other steps to protect S' information. Any other public statements regarding the trial requires prior written consent from S.

DOCUMENTS (2):
  • Study Protocol (2021-11-12): https://cdn.clinicaltrials.gov/large-docs/61/NCT04881461/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/61/NCT04881461/SAP_001.pdf